CLINICAL TRIAL: NCT03376308
Title: Evaluation of the Effect of Venous Diameter Measurement by Ultrasonography on Pain and Withdrawal Response
Acronym: VDIAMETER
Status: Completed | Type: Observational
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, SİNAN YILMAZ, Principal Investigator, Aydin Adnan Menderes University
Other Study IDs: VASCULAR DIAMETER
Record Dates: First submitted 2017-12-13; First posted 2017-12-18 (Actual); Last update posted 2017-12-19 (Actual); Status verified 2017-11

CONDITIONS: Pain; Withdrawal
Keywords: rocuronium; propofol; pain; withdrawal; venous diameter
MeSH Terms: conditions — Pain | interventions — Neurovascular Coupling

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Venous diameter measurements were made via the USG in the hand dorsum. Transverse venous diameter ≤2mm was defined group 1.
  Anesthesia induction drugs were all treated in the same order and dose. Pain score, withdrawal movement score and hemodynamic response was recorded.
  Interventions: Diagnostic Test: Pain Score; Diagnostic Test: Withdrawal movement score; Diagnostic Test: hemodynamic response
- Group 2: Venous diameter measurements were made via the USG in the hand dorsum.Transverse venous diameter >2mm was defined group 2.Anesthesia induction drugs were all treated in the same order and dose.
  Pain score, withdrawal movement score and hemodynamic response was recorded.
  Interventions: Diagnostic Test: Pain Score; Diagnostic Test: Withdrawal movement score; Diagnostic Test: hemodynamic response

INTERVENTIONS:
Diagnostic Test: Pain Score — Four poin scala 0=No Pain
  1. mild
  2. intermediate
  3. severe
Diagnostic Test: Withdrawal movement score — Withdrawal movements
  1. no movement response
  2. movement limited to the wrist
  3. movement limited to the elbow/shoulder,
  4. generalized movement response.
Diagnostic Test: hemodynamic response — Hemodynamic data were recorded in the patients taken in the operation room. (T0). Hemodynamic values (T1) measured 1 minute after administration of intravenous propofol were recorded. Hemodynamic values (T2) measured 1 minute after administration of intravenous rocuronium were recorded. Hemodynamic values (T3) measured 1 minute after administration of endotracheal intubation were recorded.

SUMMARY:
During general anesthesia, intravenous (IV) medications can disrupt the patient's comfort by causing a pain sensation or a withdrawal response in the heart. Propofol and rocuronium are among the most common causes of this condition.

In recent years, the use of ultrasonography (USG) in anesthesia has become widespread with the rapid advancement of technology. The use of the patient's head is a non invasive method.

This study is aimed to evaluate whether the size of the venous diameter assessed by ultrasonography in our study is an effect on pain and withdrawal response after drug injections.

DETAILED DESCRIPTION:
The study was conducted in patients who underwent surgical procedures under general anesthesia by obtaining consent from the Adnan Menderes University Medical Faculty Ethics Board and written consent from the patients and then being admitted to the ASA I-II age group 18-70 years of age.

Patients with peripheric vascular disease, vasculitis, rheumatologic disease, non-cooperative, under the age of 18 and over 70, ASA III and above, allergic to general anesthetic agents and refusing to participate in the study were excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

18- 70 years of ASA (American society of anesthesiology) physical status I- II who were to undergo various elective operations

Exclusion Criteria:

Rheumatologic disease Peripheric vascular disease Vasculitis Patients with chronic pain syndrome, Patients with neurologic deficits, Patients with thrombophlebitis, Patients with difficult venous access, Patients with allergy

Ages: 17 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study was conducted on 145 patients aged 17- 70 years of ASA (American Society of Anesthesiologists) physical status I- II who were to undergo various elective operations. None of the patients was premedicated before the operation. Venous diameter measurements were performed in preoperative room via USG.The patients were monitored with three derivation electrocardiogram, non- invasive arterial pressure, and pulse oximeter.
Sampling Method: Probability Sample
Enrollment: 145 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
The injection pain due to propofol | 6 month
  Pain will be recorded and graded using a 4-point scale (none, mild, moderate, or severe).

SECONDARY OUTCOMES:
The withdrawal movement due to rocuronium | 6 month
  Withdrawal movements are scored as follows: (a) no movement response, (b) movement limited to the wrist, (c)movement limited to the elbow/shoulder, or (d) generalized movement response.

CONTACTS AND LOCATIONS:
Overall Officials: Sinan Yılmaz, Principal Investigator — Aydin Adnan Menderes University
Locations (1):
- Adnan Menderes University Training and Research Hospital, Aydin, Turkey (Türkiye)